CLINICAL TRIAL: NCT01564628
Title: Data Acquisition for Optimization of Coronary Artery Disease Algorithm
Brief Title: Data Acquisition for Optimization of Coronary Artery Disease (CAD) Algorithm
Status: Completed | Type: Observational
Sponsor: Acarix (Industry)
Responsible Party: Sponsor
Other Study IDs: AC003-SH
Record Dates: First submitted 2012-03-21; First posted 2012-03-28 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: Population from 2 sites, sequential design with all patients undergoing CADScor1 intervention followed by the diagnostic testing the patients were referred to (procedure done according to standard of care and not part of study; computerized tomographic angiography (CTA) and, if relevant, coronary angiography (CAG) at Site 1 and CAG at site 2).
  Interventions: Device: CADScor1

INTERVENTIONS:
Device: CADScor1 — Acoustic recording

SUMMARY:
The purpose of the study is to optimize an already existing algorithm for diagnosing atherosclerosis of the coronary arteries (CAD, Coronary Artery Disease).

DETAILED DESCRIPTION:
Acoustic information from the heart is obtained from patients referred to examination for Coronary Artery Disease. The acoustic signals are evaluated as indicators for CAD.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Referred to diagnostically Ca-CT, CT scan and/or CAG examination due to suspicion of coronary artery disease
* Subjects condition must be stable and the subject must not be referred due to suspicion of acute coronary syndrome
* Subject is willing to adhere to the study procedure
* Has signed the informed consent form and authorization to registration and publication of health information

Exclusion Criteria:

* Has acute coronary syndrome or stroke
* Arterial fibrillation
* Known severe arrhythmia or resting heart rate above 85 bpm
* Known diastolic murmurs due to heart valve disease
* Has had a previous by-pass operation, open chest surgery, donor heart or mechanical heart
* Reduced ejection fraction < 50%
* Inability to understand or adhere to instructions for acoustic Data-acquisition (i.e. subject not able to hold breath due to KOL or asthma)
* Inability to perform CT-angio and/or subsequent CAG
* In active treatment for any cancer
* In active treatment for immunosuppression after transplantation
* Established or pursuing pregnancy or breast feeding
* Has damaged skin on the spot where the patch is placed during the recordings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to examination for Coronary Artery Disease
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morten Bøttcher, MD, Principal Investigator — University Hospital of Aarhus, Skejby
Locations (1):
- University Hospital of Aarhus, Skejby, Aarhus N, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Site 1A Population - CAD-score/CTA/CAG: Site 1A study population. Subject to CAD-score, CTA and, if relevant, CAG investigation.
- Site 2 Population - CAD-score/CAG: Site 2 study population. Subject to CAD-score and CAG investigation
- Site 1B Population - CAD-score/CTA/CAG: Site 1B study population. Subject to CAD-score, CTA and, if relevant, CAG investigation
Period: Overall Study
Arm/Group | Site 1A Population - CAD-score/CTA/CAG | Site 2 Population - CAD-score/CAG | Site 1B Population - CAD-score/CTA/CAG
Started | 185 | 58 | 63
Completed | 181 | 56 | 61
Not Completed | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Population: PP population.
Arm/Group | All Study Participants
Number analyzed (Participants) | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 160
Region of Enrollment [Number; unit: participants]
  Denmark | 298

OUTCOME MEASURES:

1. Primary Outcome: The Area Under the Receiver Operating Characteristic Curve of the CAD-score to Separate CAD From Non-CAD Patients.
Description: Cardiac noise marker (CAD-score) ability to separate CAD from non-CAD patients is estimated as the area under the receiver operating characteristic curve.
  The area under the receiver operating characteristic curve is plottet as sensitivity versus 1-specificity as a function of different CAD-score cut-off values.
  The area under the receiver operating characteristic curve is on a scale from 0-100%, the higher value means a better separation of CAD from non-CAD patients.
  CAD and non-CAD patients are defined by the CTA and CAG evaluations.
Time Frame: Heart sound recordings measured on testday (25 minutes study period)
Population: Per protocol analysis
Measure: Mean (95% Confidence Interval); unit: percentage of 100
Arm/Group | All Study Participants
Number analyzed (Participants) | 298
percentage of 100 | 73.4 [66.2 to 80.0]

ADVERSE EVENTS:
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/298
Serious Adverse Events (participants affected / at risk) | 0/298
Other Adverse Events (participants affected / at risk) | 0/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less